CLINICAL TRIAL: NCT04558398
Title: The Impact of Short-term Exercise Programs on Mitochondrial Activity in Colorectal and Prostate Cancer Patients.
Brief Title: Impact of Exercise on Mitochondria in Cancer Patients.
Acronym: ICCE-Mito
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21018
Record Dates: First submitted 2020-02-14; First posted 2020-09-22 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer; Colorectal Cancer
Keywords: Mitochondrial activity; Resistance exercise training; High-intensity interval training
MeSH Terms: conditions — Prostatic Neoplasms; Colorectal Neoplasms | interventions — Resistance Training; High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants will all receive baseline assessments of their mitochondrial function, muscle mass and functional assessments.
  Participants with both cancer types (Prostate and colorectal) will be randomly allocated to either Resistance based or high-intensity interval training based home exercises for 4 weeks prior to their planned surgical date.
  Participants will then all be re-assessed on the day of their planned surgical procedure.
Masking Description: Due to the nature of the exercise interventions, there will be no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise training group (Experimental): Participants randomized to this arm will engage in a 4-week home-based training program with anticipated 12 sessions (3 per week) with participants required to attend a minimum of 9 sessions.
  Interventions: Other: Resistance exercise training
- High-intensity interval training group (Experimental): Participants randomized to this arm will engage in a 4-week home-based training program with anticipated 12 sessions (3 per week) with participants required to attend a minimum of 9 sessions.
  Interventions: Other: High-intensity interval training

INTERVENTIONS:
Other: Resistance exercise training — Each session will be performed at home, with resistance bands used to provide resistance. Participants will be guided to increase the resistance if over 15 repetitions can be performed prior to fatigue. Weekly contact will be made with participants to encourage participation and to guide the exercise.
  Each session will include:
  2 min warm-up jogging on the spot
  2 sets of 12-15 repetitions of:
  Squats
  Hip flexion
  Hip extension
  Hip abduction
  Seated row
  Bench press
  Lateral raises
  2 min jogging on the spot cooldown.
  Arms: Resistance exercise training group
Other: High-intensity interval training — Each session will include:
  * 2 min warm-up: jogging on the spot
  * Each of the following exercises performed for 60seconds, interspaced by 90 seconds rest
    * Star jumps
    * Standing squats
    * On-the-spot sprints
    * Standing squats
    * Star jumps
  * 2 min cool-down: jogging on the spot
  Participants will be contacted weekly to encourage participation and to guide the exercise
  Arms: High-intensity interval training group

SUMMARY:
The aim is to investigate the impact of prostate and colorectal cancer on mitochondrial quantity and quality along with muscle mass and function and whether this can be modified through the use of a home-based short-term exercise training program.

The investigators aim to recruit participants awaiting curative surgery for colorectal and prostate cancer and to assess the variation in baseline mitochondrial activity between them.

Participants from both cancer types will then carry out a 4 week home exercise program, this will be randomly allocated to either resistance-based or high-intensity interval training based. Participants will then be re-assessed on the day of their planned surgical procedure to assess the changes effected by the training program.

The investigators hypothesize that there will be variation in mitochondrial activity linked to muscle mass across the two cancer types and that home-based exercise programs have the ability to improve mitochondrial activity along with muscle mass.

DETAILED DESCRIPTION:
Participants will be recruited from surgical outpatient clinics following an initial introduction to the trial by their clinical team. At this point, participants will be provided with a participant information sheet. Contact details will be provided on the information sheet to enable potential participants to arrange a screening visit. The screening visit would entail a detailed description of all study elements and addressing any questions prior to gaining written consent. Once the patient provides written informed consent, they will undergo a full cardiovascular examination by a medically qualified research team member and will have a set of screening bloods taken.

D2O Instructions 24 hours prior to the study day, participants will be asked to consume a stable isotope tracer drink (D2O) at a 3 ml/kg priming dose at home. Participants will be asked to provide saliva samples immediately prior to D2O consumption and a further sample 2-hours post-consumption. Participants will be provided with written instructions, the tracer drinks, and collection receptacles at their screening visit or via postal delivery for them to collect these samples at home. Participants will also be provided with a smaller maintenance dose (1.5ml/kg) to maintain D2O enrichment throughout the training program. This will need to be consumed once per week, with saliva collected immediately prior to, and 2-hours post-consumption each week - again, all materials and written instructions will be provided.

Pre-Exercise study day Participants will attend the University of Nottingham Graduate Entry Medical School at the Royal Derby hospital for an assessment visit prior to the commencement of their training protocol. Participants will be asked to arrive starved from 03:00 of the day, this is to match the nil-by-mouth rules required for their surgical procedure to ensure that all assessments are performed on the same fed-state. On arrival, they will undergo a limited number of physical function assessments (including time up and go, handgrip strength, and the short performance physical battery test).

Followed by the Ruffier test to provide an estimated cardiopulmonary fitness[14]. The ruffier test is performed by the participant resting for 5 minutes (lying down) then taking note of the resting heart rate. The participant then performs up to 30 standing squats within 45seconds, with a heart rate taken immediately upon completion. The participant then lies back down for 2 minutes with further heart rate measurement. This allows us to calculate the Ruffier Dicksons index which provides an estimated cardiopulmonary fitness[15].

Ruffier Dickson index (RDI): ((P1-70)+ 2(P2-P0))/10 Where P0 is 15 s average resting HR, in our case, from 3 min 45 s to 4 min, P1 is the maximum HR recorded during the first 15 s of recovery, and P2 is the 15 s average after the 1st minute of recovery, that is from 1 min and 00 s and 1 min and 15 s.

An ultrasound scan of the thigh to assess muscle architecture will then be performed.

A muscle biopsy will be taken from the mid-belly of m. vastus lateralis using a conchotome biopsy technique. Biopsies will be taken by medically qualified doctors trained and experienced in this procedure. The procedure will be performed under aseptic conditions. After local anesthetic; a 5-10mm incision will be made in the skin and underlying fascia and a sample of muscle will be taken (approximately 150mg). Direct pressure will be applied to achieve hemostasis. A single absorbable suture will be placed to allow skin apposition and healing. A sterile dressing and compression bandage will be applied to remain in place for the duration of the day. The suture will dissolve around 7-10 days after the biopsy was taken. The biopsy sample will be assessed using an Oroboros respirometer for the primary endpoint of mitochondrial activity, analysed by western blotting, PCR and immunohistochemistry to determine cell signalling and gene expression.

Participants will then be provided with a complimentary snack, and asked to complete quality of life questionnaires (EQ-5D and IPAQ). Participants will be randomly allocated to either the training arm of the study or to routine care at this point. The training regimen will then be demonstrated to them with time allowed for questions regarding the training regimen. This will conclude this study day.

Training program:

All exercise training will take place in the participants own home. With a documentation pack provided to participants to guide exercise and for participants to log their workouts.

Participants will be asked to perform 3 workouts per week over the 4-week period (12 workouts in total) with each workout estimated to take 30 minutes maximum.

Participants randomly allocated to the resistance group will be provided with a set of resistance bands to provide resistance to their workout.

As well as the education session provided at the pre-exercise study day, participants will be contacted weekly via telephone or video call to provide support, encourage participation, answer any difficulties participants maybe experiencing, and to ensure no adverse symptoms are being experienced. A video will be recorded of a member of the research team performing the exercise regimen to enable participants to watch from home.

For participants in the RET arm, the session will include:

2 min warm-up jogging on the spot 2 sets of 12-15 repetitions of: Squats Hip flexion Hip extension Hip abduction Seated row Bench press Lateral raises 2 min jogging on the spot cooldown.

Each exercise will be separated by 1-minute rest, with participants encouraged to workout to mild fatigue on their final repetition in each set. If able to perform more than the allocated maximum of 15 repetitions prior to fatigue, then participants will be informed to increase the resistance by using a tougher resistance band.

For participants in the HIIT arm, the session will include:

2 min warm-up: jogging on the spot Each of the following exercises performed for 60seconds, interspaced by 90 seconds rest Star jumps Standing squats On-the-spot sprints Standing squats Star jumps 2 min cool-down: jogging on the spot

Our research group has conducted many similar exercise regimes of this intensity to subjects in the anticipated age-range without incident. Participants will be advised to terminate exercise training immediately if experiencing:

Chest pain or tightness Faintness Sudden pallor Loss of co-ordination Confusion Dizziness Palpitations Sudden breathlessness

Should any participant experience these effects during any session, they will be advised to seek urgent medical attention and will be withdrawn from the study for safety purposes.

Day of surgery study day All participants will attend for their operations fasted as per the clinical teams' instructions, this is to be starved 6-hours prior to anticipated surgical start time, in line with anesthetic guidelines. Participants will be met by a member of the research team on their arrival, who will perform the following assessments during the time prior to their surgery. Participants will first have an ultrasound scan of the thigh to assess muscle architecture. Following this, participants will be asked to complete a quality-of-life questionnaire (EQ-5D) and a self-administered short-form international physical activity questionnaire (IPAQ). The sputum samples collected at home will be received from the participants by a researcher. Participants will then perform physical function assessments to determine muscle function, including the timed-up-and-go test, and the short performance physical battery test, and the ruffier test to provide an estimated VO2. These assessments will all be completed by a member of the research team prior to the participant being taken to theatre and will not delay a participant's surgical start time, nor will it require participants to arrive earlier than patients not undertaking the study.

Once the participant has been anesthetized for their planned surgical procedure, a member of the research team perform venipuncture to gather samples for analysis of myokine expression, this will be followed by a single muscle biopsy. The muscle biopsy will be taken from the mid belly of m. vastus lateralis using the conchotome biopsy technique as previously described.

Day 21-28 post-surgery Participants will be contacted by postal survey and asked to complete a further EQ-5D and IPAQ questionnaire, along with a study feedback questionnaire to ascertain participants views on the study and their exercise program.

As detailed above, in addition to their normal treatments, patients will potentially undergo the following invasive or potentially harmful tests from involvement in the study (risks outlined in Risk section): three blood tests and 2 muscle biopsies.

ELIGIBILITY:
Inclusion criteria

1. Aged 50 years and over (no upper age limit)
2. Male patients
3. Histologically confirmed malignancy, radiologically or direct visualisation leading to high clinical suspicion of cancer with planned surgical resection as treatment option (prostate or colorectal).
4. Sufficient mobility to be able to complete a home-based exercise program
5. Capacity to give informed and written consent
6. Ability to travel to the RDH to complete the assessment session

Exclusion criteria

1. Current participation in a formal exercise regime
2. Inability to complete exercise training
3. Inadequate level of the English language to be able to provide consent
4. A BMI <16.5 or >35 kg/m2
5. Active cardiovascular disease:

   1. Uncontrolled hypertension (BP > 160/100)
   2. Angina
   3. Heart failure (class III/IV)
   4. Significant arrhythmia
   5. Right to left cardiac shunt
   6. Recent cardiac event
6. Taking beta-adrenergic blocking agents
7. Cerebrovascular disease:

   g. Previous stroke h. Aneurysm (large vessel or intracranial) i. Epilepsy
8. Respiratory disease including:

   j. Pulmonary hypertension k. Significant COPD l. Uncontrolled asthma
9. Clotting dysfunction or current use of anticoagulants (eg Warfarin/Clopidogrel/ Rivaroxaban)
10. Significant musculoskeletal or neurological disorders
11. Female patients
12. Those requiring or receiving neoadjuvant chemotherapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial activity across 2 cancer types | Assessed at initial baseline study day across cancer types
  Mitochondrial oxidative phosphorylation capacity between colorectal and prostate cancer.
  Mitochondrial oxidative phosphorylation capacity will be measured according to oxygen consumption determined by the use of a high-definition respirometer. This will then be compared across cancer types and expressed as a ratio of maximal consumption.
Mitochondrial activity change with a short-term home-based exercise program | Assessed over the 4-weeks prior to planned surgical resection
  The effect of either a resistance exercise-based and high-intensity interval training-based home-based training program on mitochondrial function.
  Mitochondrial oxidative phosphorylation capacity will be measured according to oxygen consumption determined by the use of a high-definition respirometer. The changes seen throughout the treatment will then be expressed as a percentage in order to express the changes seen from the baseline.
The altered response to training - type between cancer type. | 4-weeks
  The differing responses between cancer type to the short-term exercise training.
  Mitochondrial oxidative phosphorylation capacity will be measured according to oxygen consumption determined by the use of a high-definition respirometer. The changes caused by the training regimen will then be expressed as a percentage in order to express the changes seen from the baseline, and in order to allow comparison between cancer type.

SECONDARY OUTCOMES:
The difference in muscle-function compared between cancer types, and its change throughout a short-term exercise program. | 4-weeks
  As assessed using the short performance physical battery tests. This is a well-established measure of lower extremity physical function, giving a maximal numerary score out of 12 allowing comparison between cancer-types and throughout exercise regimen.
The effect of cancer types and exercise on myokine expression. | 4-weeks
  Myokines planned to be analysed: Interleukin - 6, Tumour necrosis factor- alpha, and transforming growth factor beta.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Lund, MD MBBS, Principal Investigator — Nottingham University
Locations (1):
- Thomas Smart, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No